CLINICAL TRIAL: NCT04091074
Title: Safety and Effectiveness of Ticagrelor in Patients Undergoing Carotid Stenting
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Ibrahim Aboelfath Ibrahim, Osama Ibrahim Aboelfath Ibrahim, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ticagrelor in carotid stenting
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin + ticagrelor before carotid stenting (Active Comparator): patients undergoing carotid stenting take aspirin 150 mg + ticagrelor 90mg for 15 days before carotid stenting
  Interventions: Drug: Ticagrelor; Procedure: Carotid stenting
- aspirin + clopidogrel before carotid stenting (Active Comparator): patients undergoing carotid stenting take aspirin 150 mg + clopidogrel 75 mg for 15 days before carotid stenting
  Interventions: Drug: Clopidogrel; Procedure: Carotid stenting

INTERVENTIONS:
Drug: Ticagrelor — Half of patients undergoing carotid stenting take ticagrelor+aspirin
  Arms: aspirin + ticagrelor before carotid stenting
Drug: Clopidogrel — Other half ofpatients undergoing carotid stenting take clopidogrel+aspirin
  Arms: aspirin + clopidogrel before carotid stenting
Procedure: Carotid stenting — Patients with carotid stenosis will undergo carotid stenting

SUMMARY:
patients undergoing carotid stenting take dual anti platelet therapy to prevent thrombotic complications usually used drugs are aspirin plus clopidogrel but there are patients not respond so ticagrelor may be an effective and safe alternative

ELIGIBILITY:
Inclusion Criteria:

1. Ischemis stroke of both sex.
2. More than 18 years.
3. Accepting all study requirements.

Exclusion Criteria:

1. Refuse to comply with all study requirements.
2. bleeding tendency or liver diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
compare efficacy of ticagrelor and clopidogrel in patients undergoing carotid stenting | 15 days before carotid stenting
  patients undergoing carotid stenting are divided into 2 groups comparing efficacy of ticagrelor and clopidogrel
Compare safety of ticagrelor and clopidogrel in patients undergoing carotid stenting | 15 days before carotid stenting
  Patients undergoing carotid stenting are divided into two groups comparing safety of ticagrelor and clopidogrel

SECONDARY OUTCOMES:
Pattern of carotid stenosis | 1 year
  Incidence of carotid stenosis in patients come to Assiut university hospitals